CLINICAL TRIAL: NCT02782442
Title: Cognitive Training Delivered Remotely to Individuals With Psychosis
Brief Title: Cognitive Training Delivered Remotely to Individuals With Psychosis (ROAM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2016-24813
Record Dates: First submitted 2016-03-14; First posted 2016-05-25 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Treatment; Active Control; Schizophrenia; Psychosis; Schizoaffective Disorder; Psychotic Depression; Psychotic Mood Disorders; Psychotic Disorders; Psychotic Episode; Cognitive Impairment
Keywords: Cognitive Training; Motivation Enhancement
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Affective Disorders, Psychotic; Cognitive Dysfunction | interventions — PRIME protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Cognitive Training & PRIME (Experimental): Structured cognitive training consists of social cognition and auditory exercises.
  Interventions: Behavioral: Structured Cognitive Training & PRIME
- Computer Games Control & PRIME (Active Comparator): Computer games control condition comes in the official PositScience wrapper.
  Interventions: Behavioral: Computer Games Control & PRIME

INTERVENTIONS:
Behavioral: Structured Cognitive Training & PRIME — The treatment condition-- 30-35 hours of CT over 16 weeks (~2 hours per week) is a structured program of 20 hours of auditory processing exercises followed by 10 hours of social cognition exercises, combined with the personalized PRIME coaching application
  Arms: Structured Cognitive Training & PRIME
Behavioral: Computer Games Control & PRIME — Computer games control condition which comes in the official PositScience wrapper. 30-35 hours of games over 16 weeks (~2 hours per week), combined with the personalized PRIME coaching application.
  Arms: Computer Games Control & PRIME

SUMMARY:
Primary study:

This study is a single-site, double-blind, randomized, controlled clinical trial to compare an evidence-based structured program of 30-35 hours of on-line cognitive and social cognitive training exercises performed over 16 weeks (~2 hours per week), delivered with an innovative digital app which provides users with a motivation coach to set personalized goals and with secure social networking for peer support, "PRIME" ; vs. 2) A control condition of computer games, encouraged at ~2 hours per week over 16 weeks, delivered with "PRIME".

Unblinded Cognitive Training Sub-Study:

Participants who were randomized to the computer games arm of the trial may be offered access to the active cognitive training at the end of their 6 month follow up appointments, if they still meet inclusion criteria.

PRIME Super Users Sub-Study:

Participants who have provided all follow up data to the initial study, including those who are currently enrolled in the Unblinded Cognitive Training sub-study, may be offered continued participation in the PRIME community as super-users.

DETAILED DESCRIPTION:
Primary study:

The purpose of this study is to use remote methods and scalable interactive neurotechnology to generate important data on the potential for remote targeted cognitive treatment in people with psychosis. We will perform a double-blind RCT in 120 participants with psychosis, comparing: 1) An evidence-based structured program of 30-35 hours of on-line cognitive and social cognitive training exercises (CT) performed over 16 weeks (~2 hours per week), delivered with an innovative digital app which provides users with a motivation coach to set personalized goals and with secure social networking for peer support, "PRIME"; vs. 2) A control condition of computer games, encouraged at ~2 hours per week over 16 weeks, delivered with "PRIME" . Both conditions will be administered using personal smartphone devices and computers and all procedures will be conducted remotely, including on-line recruitment in locations all over the world. Using both per protocol and intent-to-treat analyses, we will determine clinical, cognitive, and functional effects after the intervention using operationalized assessments delivered remotely, and will determine their relationship to functional outcome measures at 6-month follow-up.

Both the active condition and the control condition will be provided through identical web portals designed for the study at no charge by Brain HQ (Posit Science, Inc.). PRIME, the personalized motivation coaching and social networking app, has been designed and developed by co-investigator Dr. Schlosser, supported by UCSF and NIMH. We will recruit a total of 204 subjects with psychosis to be stratified by age (18-40, 40-60) and education (< 14 years, >14 years) and randomly assigned to one of the two conditions.

Unblinded Cognitive Training Sub-Study:

During the debrief, participants will be asked if they would like to continue participating in the study and receive active cognitive training. If the participant agrees, they will sign a new consent form which covers the details of the next portion of the study. The data from their 6 month follow up appointment will be counted as their baseline data to reduce participant burden. They will start immediately with cognitive training and will continue through the 6 month follow up appointments, as above. Additionally, participants who enter into this study may be offered simultaneous participation in the PRIME Super Users sub-study (see below).

PRIME Super Users Sub-study:

As a super-user, PRIME members are asked to take on a peer-mentorship role in the community and maintain a certain level of activity within the application. Before offering participation in the sub-study, the study team will perform a case review to determine if PRIME would be beneficial to the individual, that they appear able to fulfill the role of a peer mentor, that they are likely to be consistently active within the community, and they are able to adhere to the PRIME code of conduct. Participants will sign informed consent before rejoining the community.

As super-users, participants will be asked to be active members within the community and to maintain activity of once a week, on average. Participants will be asked to notify study staff if they anticipate or experience any extended absences from the app for any reason so their access to the community will not be revoked. Super-users will participate in the community by making posts, sharing moments, and commenting on the posts of other community members (including ROAM participants, Super-Users, and coaches). They are encouraged to share stories from their experiences and offer advice to other users for making and achieving goals, dealing with symptoms, and improving quality of life.

ELIGIBILITY:
Inclusion Criteria for the primary study:

1. SCID confirmed clinical diagnosis of the following: schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis NOS, major depressive disorder with psychotic features, or bipolar disorder with psychotic features.
2. Good general physical health.
3. Between the ages of 18 and 60 years old at the time of screening.
4. Be fluent in spoken and written English, in that the participant learned to speak English before the age of 12 or is able to demonstrate fluency in conversation with study staff, or through English language exams, such as TOEFL, or English language courses
5. No neurological disorder.
6. Have an outpatient status of at least 1 month prior to participation.
7. Been on a stable dose of psychiatric medications for at least one month prior to participation (may include no medication).
8. Have a personal smartphone
9. Have access to a computer.
10. No prior cognitive training experience within the past 3 years.
11. Pregnant women may participate in this study.

Inclusion Criteria for Unblinded Cognitive Training Sub-Study:

1. Continues to meet inclusion criteria for ROAM (except for access to smart phone)
2. Has completed 6 month assessments for ROAM
3. Was randomized to the control condition (computer games) and did not receive active cognitive training.

Inclusion Criteria for the PRIME Super Users sub-study:

1. Has participated in the 6 month assessments for ROAM
2. Has shown adequate participation in PRIME during the ROAM study (e.g., active in PRIME community once a week on average)
3. Has adhered to the PRIME App and Study Rules
4. Is clinically stable and, in the opinion of the study staff and PRIME coaches, does not pose a risk to themselves or the PRIME community by continuing participation.
5. Is capable of participating in the PRIME community independently with minimal support from study staff or PRIME coaches.
6. Had a positive experience with the PRIME community and appears to be capable of positively contributing to the community.

Exclusion criteria for all studies:

1. We will exclude participants with a history of severe substance abuse in the past 3 months determined by DSM criteria.
2. Subject is unable to demostrate adequate decisional capacity, in the judgment of the consenting staff member, to make a choice about participating in the research study.
3. Anyone who does not meet the aforementioned inclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Penn Computerized Neurocognitive Battery MATRICS Protocol (Penn CNB) | Baseline, Immediately after Intervention, 6 Month Follow-Up
  A series of computerized tests administered remotely that measure performance accuracy and speed on specific neurocognitive domains
Change in Abbreviated Quality of Life Scale (aQLS) | Baseline, Immediately after Intervention, 6 Month Follow-Up
  A semi-structured interview which evaluates psychosocial functional outcome. Item scores range from 0 to 6 with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Change in Behavioral Inhibition System/Behavioral Activation System (BIS-BAS) | Baseline, Immediately after Interviention, 6 Month Follow-Up
  A self-report measure of motivation examining both motivation to avoid aversive outcomes and motivation to approach goal-oriented outcomes. Item scores range from 1 to 4. BIS: lower scores indicate more behavioral inhibition (a worse outcome). BAS: lower scores indicate more behavioral activation (a better outcome).
Change in Motivation and Pleasure Scale (MAP-SR) | Baseline, Immediately after Intervention, 6 Month Follow-Up
  A self-report measure of the severity of negative symptoms. Item scores range from 0 to 4 with higher scores indicating a better outcome.
Change in Role Functioning Scale (RFS) | Baseline, Immediately after Intervention, 6 Month Follow-Up
  A measure of the level of functioning in four domains: working productivity, independent living and self care, family network relationships, and immediate social network relationships. Item scores range from 1 to 7 with higher scores indicating a better outcome.
Change in Quick Scale for the Assessment of Negative Symptoms/Quick Scale for the Assessment of Positive Symptoms (Q-SANS/Q-SAPS) | Baseline, Immediately after Intervention, 6 Month Follow-Up
  A semi-structured interview assessing the severity of negative and positive symptoms of psychosis. Item scores range from 0 to 100 with lower scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota Department of Psychiatry
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Primary outcome data will be shared with the NIH Data Archive in the National Database for Clinical Trials related to Mental Illness.
  De-identified data will be available for sharing with other researchers upon request. Data will not be released until 6 months after the first publication of results from this study. The protocol, consent documents, statistical analysis plan, and analytic code may be made available upon request, per PI discretion.
  In addition to the primary and secondary outcome measures listed above, there are several experimental measures which have been collected in this study. These data may also be available for sharing with other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will first be available for sharing 6 months after first publication of results. There is no planned end date to availability of data after release.
Access Criteria: Collaborators must request permission of the PI for access to the data. Additionally, any interested parties must complete a Data Use Agreement for access to the data.

REFERENCES:
- [Derived] Fisher M, Etter K, Murray A, Ghiasi N, LaCross K, Ramsay I, Currie A, Fitzpatrick K, Biagianti B, Schlosser D, Loewy R, Vinogradov S. The Effects of Remote Cognitive Training Combined With a Mobile App Intervention on Psychosis: Double-Blind Randomized Controlled Trial. J Med Internet Res. 2023 Nov 13;25:e48634. doi: 10.2196/48634. PMID 37955951